CLINICAL TRIAL: NCT00243828
Title: Assessment of the Effectivity of Total-face Mask for Noninvasive Ventilation During Acute Respiratory Failure: a Randomized Controlled Trial.
Brief Title: Assessment of the Effectivity of Total-face Mask for Noninvasive Ventilation During Acute Respiratory Failure
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Very low rate of recruitment anticipated futility of pursuing the study
Sponsor: Corporacion Parc Tauli (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEIC2005/022; AATRM 151/23/2004
Record Dates: First submitted 2005-10-24; First posted 2005-10-25 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2007-03

CONDITIONS: Respiratory Insufficiency
Keywords: Noninvasive Mechanical Ventilation; Acute Respiratory Failure; Intubation
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Total Face Mask

SUMMARY:
Total-face mask may improve the efficacy of NIV compared to conventional face mask in patients with acute respiratory failure due to enhanced tolerance and the allowance of higher airway pressure without massive leaks.MAIN OBJECTIVE: To assess, in acute respiratory failure patients, whether the total-face mask reduce the intubation rate. METHODS: 300 patients admitted in the ICU for acute respiratory failure needing continuous noninvasive mechanical ventilation. The type of mask (total-face vs. conventional face mask) will be randomized. Defined failure criteria and weaning technique will be used.

DETAILED DESCRIPTION:
HYPOTESIS: Total-face mask may improve the efficacy of NIV compared to conventional face mask in patients with acute respiratory failure due to enhanced tolerance and the allowance of higher airway pressure without massive leaks.OBJECTIVES: To assess, in acute respiratory failure patients, whether the total-face mask reduce the intubation rate. Additionally, whether it may improve mask tolerance, skin pressure damage, number of patients receiving higher pressures, or even a reduction in mortality. METHODS: 300 patients admitted in the ICU for acute respiratory failure needing continuous noninvasive mechanical ventilation. The type of mask (total-face vs. conventional face mask) will be randomized. PEEp will be titrated to the best oxygenation and IPAP up to reduce dyspnea and respiratory frequency, with the limits at clinical tolerance and massive leaks. Defined failure criteria and weaning technique will be used. Data to record include clinical parameters and mortality risk score (SAPS II), and physiologic response to NIV (either subjective and objective), technique failures and outcome. EXPECTED RESULTS: The study has been powered to detect a 30% relative improvement in intubation rate from a 35% baseline incidence of intubation in the conventional group.

ELIGIBILITY:
Inclusion Criteria:

* Acute Hypoxemia:PaO2/FiO2 lower than 200 mmHg
* Respiratory rate greater than 30 breaths/min

Exclusion Criteria:

* cardiogenic lung edema
* COPD exacerbation
* Low level of consciousness (GCS < 13)
* Hemodynamic instability
* Facial damage
* Do-not-intubate orders
* Lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2005-11; Primary Completion 2007-09 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Intubation rate

SECONDARY OUTCOMES:
Hospital survival

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Fernandez, MD, PhD, Study Director — Corporacion Parc Tauli
Locations (1):
- Hospital de Sabadell, Sabadell, Barcelona, Spain